CLINICAL TRIAL: NCT01776164
Title: Early and Longitudinal Assessment of Neurodegeneration in the Brain and Spinal Cord in Friedreich's Ataxia
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: Bob Allison Ataxia Research Center (Unknown); Friedreich's Ataxia Research Alliance (Other)
Responsible Party: Sponsor
Other Study IDs: 1210M22281
Record Dates: First submitted 2013-01-14; First posted 2013-01-28 (Estimated); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Friedreich Ataxia
Keywords: Friedreich; ataxia; FRDA; FA; recessive; neurodegenerative; cerebellum
MeSH Terms: conditions — Friedreich Ataxia; Ataxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patient with FRDA: Patients affected by Friedreich's ataxia
- Healthy controls: Healthy volunteers age- and gender-matched with no neurological disease identified.

SUMMARY:
Friedreich's ataxia is characterized by progressive alterations in the function of the cerebellum accompanied by an atrophy of the spinal cord. Although the genetic defect responsible for the disease has been identified more than 15 years ago, objective markers of the pathologic process (i.e., biomarkers) that would allow measuring the effects of potential therapies are still lacking. Moreover, it is still unclear how the malfunction of the cerebellum affects the rest of the brain, and understanding the connectivity and neurochemistry of the central nervous system might yield new insights in the understanding of the disease, in addition to providing potential markers.

To address these needs, the investigators aim at utilizing the capabilities of Magnetic Resonance Imaging (MRI) and Spectroscopy (MRS). Using techniques called Diffusion Imaging, resting-state functional MRI, and Proton Spectroscopy (1H MRS), the investigators propose to determine the differences in the connectivity and neurochemistry of the spinal cord and the brain between patients affected by Friedreich's ataxia and healthy controls. The investigators plan on imaging both patients and control subjects using a 3T magnet, a system that although not yet available in all medical facilities, is becoming standard in most hospitals and clinics. The first aim is to scan patients already scanned last year (12-month follow-up). The second aim is to scan patients at an early stage of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Genetic diagnosis of Friedreich's ataxia for patient volunteers with GAA repeat expansion number
* Absence of neurological conditions for control volunteers
* Control volunteers will be age-, race-, and gender-matched to the patients

Exclusion Criteria:

* Claustrophobia
* Smoking
* Diabetes
* Pregnancy or lactation
* Weight over 300 lbs
* Presence of a pacemaker or any paramagnetic object in the body
* Severe scoliosis

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Friedreich's ataxia at the early stage of the disease (e.g. ambulatory and not wheelchair bound and no to early cardiomyopathy) Age- and gender-matched healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2013-01; Primary Completion 2022-02-08 (Actual); Study Completion 2022-02-08 (Actual)

PRIMARY OUTCOMES:
Difference in connectivity (apparent coefficient of diffusion, fractional anisotropy, radial and axial diffusivity), anatomy (cortical thickness, volumetry analysis) and biochemistry (metabolite concentrations) between patients and controls | 1 year
  The investigators will look at the differences between patients and controls. This is observational, not interventional.
  The fractional anisotropy (FA) is a scalar value. The apparent coefficient of diffusion, radial and axial diffusivity are measured in mm2/s. The metabolite concentrations in the brain are in the order of µg/ g wet tissue weight. Cortical thickness is measured in mm.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Gilles Henry, Ph.D., Principal Investigator — University of Minnesota; Christophe Lenglet, Ph.D, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States